CLINICAL TRIAL: NCT04382807
Title: Internet-delivered Group Counseling for Chronic Tinnitus
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Laure Jacquemin, Principal Investigator, University Hospital, Antwerp
Other Study IDs: 17/43/481
Record Dates: First submitted 2020-05-05; First posted 2020-05-11 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Tinnitus, Subjective
Keywords: tinnitus treatment; delivery method; psycho-educational counseling; internet-based
MeSH Terms: conditions — Tinnitus | interventions — Counseling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjective, chronic tinnitus: Tinnitus patients who received internet-based psycho-educational counseling
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Counseling — Online delivered group counseling session, providing insights into the tinnitus symptoms

SUMMARY:
In the treatment of chronic tinnitus, psycho-education plays an import role to provide more insights into the symptoms of tinnitus. However, the need for e-health is increasing. As such, it is important to investigate if these psycho-education sessions can be delivered online, with the same efficacy compared to the traditional face-to-face delivery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with subjective, chronic tinnitus

Exclusion Criteria:

* Enrollment in other tinnitus treatments simultaneously at the time of the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjective, chronic tinnitus patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Tinnitus Functional Index (TFI) | before intervention, 3 months follow-up
  Tinnitus severity self-report questionnaire, ranging from 0-100 with a higher score representing a more severe tinnitus.

SECONDARY OUTCOMES:
Change in Visual Analogue scale (VAS) for tinnitus loudness | before intervention, 3 months follow-up
  Visual analogue scale measuring tinnitus loudness from 0-100, with a higher score representing a louder tinnitus
Change in Hospital Anxiety and Depression Scale (HADS) | before intervention, 3 months follow-up
  Self-report questionnaire concerning anxiety and depression symptoms, ranging from 0-21 for each subscale. A result greater than 8 suggests the presence of a depression and/or anxiety disorder.
Change in Hyperacusis Questionnaire (HQ) | before intervention, 3 months follow-up
  Hyperacusis severity self-report questionnaire, ranging from 0-42 with a higher score representing a higher sensitivity to sounds. A score of 28 is the cut-off for auditory hypersensitivity.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided